CLINICAL TRIAL: NCT00824876
Title: Orthostatic Tolerance in Mamma Cancer Patients After Anaesthesia
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: OT after mastectomy
Record Dates: First submitted 2009-01-13; First posted 2009-01-19 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: Mammae cancer patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to investigate the effect of anaesthesia, on the ability to maintain upright posture immediately after surgery in mamma cancer patients.

The investigators hypothesis is, that a standard anaesthesia does not effect the ability to maintain upright posture right after surgery.

DETAILED DESCRIPTION:
It is known, that patients undergoing major surgery have problems maintaining upright posture after major surgery. This can be due to fall in bloodpressure, with symptoms like dizziness, nausea/vomiting and fainting.

With this investigation, we want to prove that anaesthesia is not the decisive factor, in patients ability to maintain upright posture after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients having performed elective breast surgery
* Age between 18 and 70 years
* Patients who have given written consent to participate in the project after haven completely understood the contents and limitations of the protocol

Exclusion Criteria:

* Patients who do not understand or speak Danish
* Patients who have not signed the informed consent or the written authority pre-medication, except 1g paracetamol
* ASA > II
* Pregnant or breastfeeding
* Known to have Renal disease
* Known to have Psychiatric disorder (not considering the use of SSRI antidepressive)
* Need for crash induction or prone position
* Oesophageal varicoses
* Necrosis or cancer in: Mouth, Pharynx, Larynx or Oesophagus
* Coarctation or aneurism in the proximal Aorta
* Severe bleeding disease

Ages: 18 Months to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mammasurgery patients
Sampling Method: Non-Probability Sample
Dates: Start 2009-01

PRIMARY OUTCOMES:
To investigate orthostatic function, measured by Finapress

SECONDARY OUTCOMES:
To investigate the occurrence of postsurgery nausea/vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, MD, Ph.D, Study Director — dept of surgical patophysiology
Locations (1):
- Dept of anesthesia 2041, ABD centre, Rigshospitalet, Blegdamsvej, Copenhagen, Denmark